CLINICAL TRIAL: NCT04592432
Title: Development of a Serious Game to Improve Nursing Students' Clinical Reasoning in the Context of Acute Heart Failure
Brief Title: Development of an Educational Video Game to Improve Nursing Students' Reasoning With Acute Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marc-André Maheu-Cadotte (Other)
Responsible Party: Sponsor-Investigator, Marc-André Maheu-Cadotte, Student, Université de Montréal
Organization: Université de Montréal (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CERSES-20-123-D
Record Dates: First submitted 2020-10-06; First posted 2020-10-19 (Actual); Last update posted 2021-04-28 (Actual); Status verified 2021-04

CONDITIONS: Heart Failure; Motivation
Keywords: Clinical reasoning; Intrinsic motivation; Serious gaming; Nursing education; Undergraduate education
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: The quantitative component is a two-group randomized crossover trial with 1:1 group allocation. Each participant will be randomly allocated to one of the two intervention sequences (i.e., the serious game SIGN@L-A followed by the serious game SIGN@L-B or vice versa). The randomization sequence list will be generated by an individual independent to quantitative data collection using an online program (randomizer.org). The primary investigator will not have access to this list. This individual will inform the primary investigator of participants' allocation after they have consented to be randomized, their randomization order based on the exact time they have completed the online consent form. Block randomization will be used with block sizes of six to avoid imbalances in group sizes.
Masking Description: Due to the nature of the interventions evaluated, participants cannot be blinded to group allocation. Furthermore, since the primary investigator is a PhD candidate and that this is his doctoral project, he will also not be blinded to group allocation as he will be responsible for assigning participants to one of the two intervention sequences and provide technical support, if needed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SIGN@L-A followed by SIGN@L-B (Experimental): Participants in this arm will have access to the prototype "SIGN@L-A" of the serious game for seven days. They will have access to this prototype from their personal computer and will be able to play with it whenever they want and for how long they wish during this period. After these seven days, they will have access the same way to the prototype "SIGN@L-B".
  Interventions: Other: SIGN@L-A; Other: SIGN@L-B
- SIGN@L-B followed by SIGN@L-A (Experimental): Participants in this arm will have access to the prototype "SIGN@L-B" of the serious game for seven days. They will have access to this prototype from their personal computer and will be able to play with it whenever they want and for how long they wish during this period. After these seven days, they will have access the same way to the prototype "SIGN@L-A".
  Interventions: Other: SIGN@L-A; Other: SIGN@L-B

INTERVENTIONS:
Other: SIGN@L-A — Two prototypes of a serious game were developed as part of this study. The design of these prototypes is based on the conceptual model by Alexiou and Schippers (2018) linking the instructional design of a serious game to intrinsic motivation, engagement, and learning outcomes. The design of SIGN@L-A will include all elements of the serious game instructional design proposed by these authors which are game mechanics (i.e., objectives to meet, feedback, and rewards), a narrative (i.e., a protagonist, non-playable characters, and narrative events), and aesthetics (i.e., functional and hedonic aesthetics).
Other: SIGN@L-B — The design of SIGN@L-B will include only some of these elements which are some of the game mechanics (i.e., objectives to meet, limited feedback), and a functional aesthetic.

SUMMARY:
The aim of this study is to appreciate, using quantitative and qualitative empirical methods, the contribution of an educational video game to the engagement, the motivation, and the development of nursing students' interpretation of acute heart failure patients' health condition. Two prototypes of the same educational video game have been developed. Study participants will play with both prototypes, complete online questionnaires and be interviewed by a research assistant regarding their experience with both prototypes. Study results will serve to select the most promising prototype between the two, based on its potential to support the engagement, the motivation, and the development of nursing students' interpretation of acute heart failure patients' health condition. Study results will also serve to refine the selected prototype before conducting a larger-scale efficacy trial. As such and given the small sample number of participants that is expected, it is not planned to conduct hypothesis testing.

ELIGIBILITY:
Inclusion Criteria:

* As part of a Bachelor of Nursing program, to be registered in a course in which acute heart failure concepts are a focus.

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2020-12-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Engagement with SIGN@L-A | Up to a week after being assigned to SIGN@L-A
  Measured with the French version of the User Engagement Scale - Short Form (Fontaine et al., 2019; O'Brien et al., 2018). This is a self-reported 5-level Likert -type scale (1 to 5). The overall score varies from 1 to 5 where a higher score is indicative of a greater engagement.
Engagement with SIGN@L-B | Up to a week after being assigned to SIGN@L-B
  Measured with the French version of the User Engagement Scale - Short Form (Fontaine et al., 2019; O'Brien et al., 2018). This is a self-reported 5-level Likert -type scale (1 to 5). The overall score varies from 1 to 5 where a higher score is indicative of a greater engagement.
Intrinsic motivation toward SIGN@L-A | Up to a week after being assigned to SIGN@L-A
  Measured with the corresponding subscale of the Échelle de motivation situationnelle (Guay et al., 2000). This is a self-reported 7-level Likert-type subscale (1 to 7). The overall score varies from 4 to 28 where a higher score is indicative of a greater intrinsic motivation.
Intrinsic motivation toward SIGN@L-B | Up to a week after being assigned to SIGN@L-B
  Measured with the corresponding subscale of the Échelle de motivation situationnelle (Guay et al., 2000). This is a self-reported 7-level Likert-type subscale (1 to 7). The overall score varies from 4 to 28 where a higher score is indicative of a greater intrinsic motivation.
Change in clinical reasoning in the context of acute heart failure | At baseline; up to seven days post-randomization
  Measured with an ad hoc questionnaire. Ten grids are presented to the participant. In each grid, a logical network between two highlighted elements must be developed. Each element refers to a concept related to acute heart failure. Each grid is then rated incorrect (0) or correct (1). The overall score varies from 0 to 10 where a higher score indicates a better clinical reasoning in the context of acute heart failure.
Change in clinical reasoning in the context of acute heart failure | At baseline; between seven and fourteen days post-randomization
  Measured with an ad hoc questionnaire. Ten grids are presented to the participant. In each grid, a logical network between two highlighted elements must be developed. Each element refers to a concept related to acute heart failure. Each grid is then rated incorrect (0) or correct (1). The overall score varies from 0 to 10 where a higher score indicates a better clinical reasoning in the context of acute heart failure.

SECONDARY OUTCOMES:
Time spent playing with SIGN@L-A | Up to a week after being assigned to SIGN@L-A
  Self-reported number of minutes estimated to have been spent playing.
Time spent playing with SIGN@L-B | Up to a week after being assigned to SIGN@L-B
  Self-reported number of minutes estimated to have been spent playing.
Degree to which the participant would like to play again with SIGN@L-A | Up to a week after being assigned to SIGN@L-A
  Measured with a self-reported 10-point scale (0: not at all; 10; a lot). The score varies from 0 to 10 where a higher score indicates a higher degree to which the participant would like to play again with the serious game.
Degree to which the participant would like to play again with SIGN@L-B | Up to a week after being assigned to SIGN@L-B
  Measured with a self-reported 10-point scale (0: not at all; 10; a lot). The score varies from 0 to 10 where a higher score indicates a higher degree to which the participant would like to play again with the serious game.
Favorite prototype of the serious game | Up to 14 days post-randomization
  Participants indicate on a questionnaire which prototype they preferred (SIGN@L-A or SIGN@L-B)

CONTACTS AND LOCATIONS:
Overall Officials: Marc-André Maheu-Cadotte, PhD(c), Principal Investigator — Université de Montréal; Patrick Lavoie, PhD, Study Director — Université de Montréal; Véronique Dubé, PhD, Study Director — Université de Montréal
Locations (1):
- Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Maheu-Cadotte MA, Dube V, Lavoie P. Development and Contribution of a Serious Game to Improve Nursing Students' Clinical Reasoning in Acute Heart Failure: A Multimethod Study. Comput Inform Nurs. 2023 Jun 1;41(6):410-420. doi: 10.1097/CIN.0000000000000966. PMID 36729896